CLINICAL TRIAL: NCT05030038
Title: Oral Aromatase Inhibitors Modify the Gut Microbiome Effecting Estrogen Bioavailability
Brief Title: Oral Aromatase Inhibitors Modify the Gut Microbiome
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00076577; WFBCCC 74121 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Gut microbiome; Circulating sex hormone metabolite concentrations
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * cPlasma will be divided into 250 mL aliquots and stored at -80 freezer in Cook Lab at BioTech Place. Blood metabolomics will be performed to identify microbial mediated metabolites using a non-targeted LC-MS/MS approach. Plasma will also be used to measure estradiol, estrone, and estrone-3-glucuronide by ELISA.
  * Fecal Samples will be mailed directly to CosmosID for DNA isolation and 12M read depth metagenomics sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aromatase inhibitor for breast cancer treatment: Participants will receive their standard of care for breast cancer treatment which includes an aromatase inhibitor. Pre-study assessments will be done at baseline as well as stool and blood samples at baseline, then again at 4 weeks and at 12 weeks during the course of the trial.
  Interventions: Biological: Fecal swab collection; Biological: Blood samples

INTERVENTIONS:
Biological: Fecal swab collection — Participants will collect fecal sample at home and either mail in the sample, or drop it off at the lab
Biological: Blood samples — Participants will have approximately 1 teaspoon of blood withdrawn from a vein, for research, on 2 different occasions. The total amount of blood withdrawn during the study will be approximately 2 teaspoons.

SUMMARY:
The purpose of this research is to study the bacteria in participants' gut before receiving a medicine called an aromatase inhibitor for breast cancer and after participants receive medicine for breast cancer.

DETAILED DESCRIPTION:
Primary Objective: To describe the microbiome shift of gut microbiome from baseline after 4-weeks and 12-weeks of oral aromatase inhibitor treatment.

Secondary Objective

* To correlate gut microbiome populations with circulating sex hormone metabolite concentrations at baseline and 12 weeks.
* To describe the correlation of change in the microbiome populations with change in circulating sex hormone metabolite concentrations from baseline to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis in situ or invasive breast cancer for which initiating aromatase inhibitors therapy is recommended or initiating aromatase inhibitors for risk reduction.
* ECOG performance status 0,1, 2, 3.
* Age ≥ 18 years
* HER2+ breast cancer is allowed if patients are on a monoclonal antibody therapy for which a change is not anticipated while on study (12 weeks) and they have been on the monoclonal antibody therapy for at least 4 weeks.
* Ability to read, understand and evaluate study materials and willingness to sign a written informed consent document.

Exclusion Criteria:

* Have been on antibiotics within 4 weeks of enrollment.
* Administered chemotherapy less than 4 weeks prior to enrollment.
* Hormone replacement (defined as only estrogen and/or progesterone replacement) or anti-estrogen therapy within 4 weeks of starting aromatase inhibitors
* Use of antibody drug conjugate (HER2+ breast cancer)
* Male breast cancer
* Any serious and/or unstable pre-existing medical, psychiatric, or other existing condition that would prevent compliance with the trial or consent process

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women of all races and ethnicity who meet the eligibility criteria are eligible for this trial.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Gut Microbial Levels - Fecal Swab | At baseline, 4 weeks and 12 weeks
  To describe the microbiome shift of gut microbiome from baseline after 4-weeks and 12-weeks of oral aromatase inhibitor treatment Investigators will calculate the change in gut microbial levels using paired t-tests.

SECONDARY OUTCOMES:
Change in Gut Microbial Levels - Blood Samples | At baseline and at 12 weeks
  Investigators will calculate Pearson or Spearman correlation coefficients between diversity and gut microbial levels and circulating sex hormone metabolite concentrations at baseline and at 12 weeks. Bacterial derived bioactive compounds, bile acids, and glucuronidated sex hormones will be compared by metabolomics conducted on plasma.
Change in Sex Hormone Concentrations - Blood Samples | At baseline and at 12 weeks
  Investigators will fit a model with independent variables of the value (baseline or 12 weeks), and a second variable that represents the change from baseline (will be 0 or the change at 12 weeks).
  Estrone, estrone-3-glucuronide, and estrone-3-sulfate concentrations will be measured using an ELISA assay conducted on plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Ansley, MD, Principal Investigator — Wake Forest Baptist Health Sciences
Locations (1):
- Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No